CLINICAL TRIAL: NCT00393679
Title: Evaluation of 4 Artemisinin-based Combinations for Treating Uncomplicated Malaria in African Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); East African Network for Monitoring Antimalarial Treatment (Network); Centre Muraz (Other); University of Calabar (Other); Tropical Diseases Research Centre, Zambia (Other Government); University Hospital Tuebingen (Other); Albert Schweitzer Hospital (Other); Uganda Malaria Surveillance Project (Other); Mbarara University of Science and Technology (Other); Ministry of Health, Rwanda (Other Government); University of Barcelona (Other); Centro de Investigacao em Saude de Manhica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4 ABC; IRB Antwerp: 6/40/187
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Fever; Malaria
Keywords: Children 6-59 months; P.falciparum; Haemoglobin; Informed consent; ACT
MeSH Terms: conditions — Fever; Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination; chloroguanil, dapsone drug combination; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): AS-AQ
  Interventions: Drug: amodiaquine-artesunate (ASAQ)
- 2 (Experimental): DHAPQ
  TO BE NOTED: since the batches of the study drug DHAPQ expire at the end of October 2008, and because of the unavailability of a new batch of DHAPQ from the manufacturer, the recruitment in the DHAPQ arm had to be discontinued on 30th October 2008. A formal amendment has been submitted to all the concerned ECs and competent authorities.
  Interventions: Drug: dihydroartemisinin-piperaquine (DHAPQ)
- 3 (Experimental): AL
  Interventions: Drug: artemether-lumefantrine (AL)
- 4 (Experimental): Lapdap + AS
  TO BE NOTED: following GlaxoSmithKline decision to discontinue the clinical development of the fixed-doses combination of Lapdap (Chlorproguanil-Dapsone) and artesunate, the Lapdap plus Artesunate arm was immediately discontinued in this study, on 17th February 2008. A formal amendment has been submitted to all the concerned ECs and competent authorities.The leading EC approval was obtained on 2nd June 2008.
  Interventions: Drug: Lapdap (Chlorproguanil-Dapsone) + artesunate (AS)

INTERVENTIONS:
Drug: amodiaquine-artesunate (ASAQ) — A fix-dose combination tablet containing artesunate-amodiaquine in three different dosages, to be used according to patient age and weight: 25mg/67.5mg; 50mg/135mg; 100mg/270mg
  Other Names: Coarsucam by Sanofi-Aventis
  Arms: 1
Drug: dihydroartemisinin-piperaquine (DHAPQ) — DHAPQ tablets contain either 20/160mg or 40/320mg of dihydroartemisinin (DHA) and piperaquine phosphate (PQ) respectively.
  Other Names: Artekin, Eurartekin by Sigma Tau; NOTE: batches expire on 31Oct08. Due to unavailability of new batches, recruitment in this arm was discontinued on 30Oct08.
  Arms: 2
Drug: artemether-lumefantrine (AL) — Tablets containing 20 mg of Artemether and 120 mg of Lumefantrine.
  Other Names: Coartem, Riamet by Novartis
  Arms: 3
Drug: Lapdap (Chlorproguanil-Dapsone) + artesunate (AS) — Lapdap tablets contain 15/18.75mg or 80/100mg of Chlorproguanil Hydrochloride and Dapsone, respectively. Arsumax® tablets contain 50mg Artesunate.
  TO BE NOTED: following GlaxoSmithKline decision to discontinue the clinical development of the fixed-doses combination of Lapdap (Chlorproguanil-Dapsone) and artesunate, the Lapdap plus Artesunate arm was immediately discontinued in this study, on 17th February 2008. A formal amendment has been submitted to all the concerned ECs and competent authorities.The leading EC approval was obtained on 2nd June 2008.
  Other Names: Lapdap by GSK.; Arsumax by Sanofi and Guilin.
  Arms: 4

SUMMARY:
The main objective is to compare the safety and efficacy of 4 artemisinin-based combinations (ACT) [amodiaquine-artesunate (AQ+AS), dihydroartemisinin-piperaquine (DHAPQ), artemether-lumefantrine (AL) and chlorproguanil/dapsone plus artesunate] for single and repeat treatments of uncomplicated malaria in children. Safety will be determined by registering adverse events and grading, laboratory, and vital signs evaluations. Their incidence will be compared between the different study arms.

TO BE NOTED: following GlaxoSmithKline decision to discontinue the clinical development of the fixed-doses combination of Lapdap (Chlorproguanil-Dapsone) and artesunate, the Lapdap plus Artesunate arm was immediately discontinued in this study, on 17th February 2008. A formal amendment has been submitted to all the concerned ECs and competent authorities. The leading EC approved the amendment on 2nd June 2008.

TO BE NOTED: since the batches of the study drug DHAPQ expire at the end of October 2008, and because of the unavailability of a new batch of DHAPQ from the manufacturer, the recruitment in the DHAPQ arm had to be discontinued on 30th October 2008. A formal amendment has been submitted to all the concerned ECs and competent authorities.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged between 6 months and 59 months inclusive. In the sites where CDA is tested all recruited children will be aged between 12 months and 59 months inclusive (this arm was discontinued on 17th February 2008). This criterion applies only for the recruitment in the first follow up. For the second follow up, children having been included in the first follow up are eligible, regardless of their age.
* Body weight of 5 Kg and above.
* Microscopically confirmed, monoinfection of Plasmodium falciparum (parasitaemia ≥ 2,000/μL to 200,000/μL).
* Fever (axillary temperature at ≥ 37.5°C) or history of fever in the previous 24 hours.
* Haemoglobin value ≥ 7.0 g/dl;
* Signed (or thumb-printed whenever parents/guardians are illiterate) informed consent by the parents or guardians. Note the informed consent will be asked only at recruitment and will cover the whole period of the study, including second active follow up and passive case detection.
* Parents' or guardians' willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

* Participation in any other investigational drug study (antimalarial or others) during the previous 30 days.
* Known hypersensitivity to the study drugs.
* Severe malaria.
* Danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand.
* Presence of intercurrent illness or any condition (cardiac, renal, hepatic diseases) which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study, including known G6PD deficiency.
* Severe malnutrition (defined as weight for height <70% of the median NCHS/WHO reference).
* Ongoing prophylaxis with drugs having antimalarial activity such as cotrimoxazole for the prevention of Pneumocystis carinii pneumonia in children born to HIV+ women.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4112 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PCR unadjusted treatment failure (TF28U): all treatment failures detected during the active follow up, regardless of genotyping. | Day 28
PCR adjusted treatment failure up to day 28 (TF28A): all early failures before day 14 plus the recurrent parasitaemias detected at day 14 or later and classified by genotyping as recrudescence. | Day 28

SECONDARY OUTCOMES:
PCR unadjusted treatment failure up to day 63 (TF63U): TF28U plus all cases of recurrent parasitaemia (symptomatic or asymptomatic) detected between day 29 and day 63 by passive follow up, regardless of genotyping | Day 63
PCR adjusted treatment failure for the whole period of passive surveillance (TFAPS): TF28A plus all episodes of recurrent parasitaemia identified as recrudescence by genotyping. | Day 28
Fever clearance time.
Asexual parasite clearance time.
Gametocytaemia (prevalence and density) at day 7, 14, 21 and 28 after treatment (for both active follow-ups); | 28 days
Hb changes day 3, 7, 14 and 28 (first and second follow up); | 28 days
Clinical malaria after first active follow-up; | 28 Days
Clinical malaria after second active follow-up; | Up to seven months
TF second clinical episode (D28 and D63); | 63 days
Changes in the frequency of mutations in the dihydrofolate reductase (DHFR) gene at day 0 first follow-up and day re-appearance of parasitaemia (for patients treated with CDA - NOTE that CDA arm was discontinued on 17.02.2008).
Safety profiles including significant changes in relevant laboratory values. | Up to seven months

CONTACTS AND LOCATIONS:
Overall Officials: UmbertoC D'Alessandro, MD MsC PhD, Study Director — Institute of Tropical Medicine Antwerp
Locations (8):
- Centre Muraz/IRSS, Bobo-Dioulasso, Burkina Faso
- Albert Schweitzer Hospital, Lambaréné, Gabon
- Manhiça Health Research Center, Manhiça, Mozambique
- Hospital, Calabar, Nigeria
- Mashshesha and Rukara, Kigali, Rwanda
- Uganda (2):
  - Jinja and Tororo, Kampala
  - Mbarara,, Mbarara
- Tropical Diseases Research Centre, P O Box 71769,, Ndola, Zambia

REFERENCES:
- [Background] Ravinetto RM, Talisuna A, De Crop M, van Loen H, Menten J, Van Overmeir C, Tinto H, Gonzalez R, Meremikwu M, Nabasuma C, Ngoma GM, Karema C, Adoke Y, Chaponda M, Van Geertruyden JP, D'Alessandro U. Challenges of non-commercial multicentre North-South collaborative clinical trials. Trop Med Int Health. 2013 Feb;18(2):237-41. doi: 10.1111/tmi.12036. Epub 2012 Dec 10. PMID 23217117
- [Result] Four Artemisinin-Based Combinations (4ABC) Study Group. A head-to-head comparison of four artemisinin-based combinations for treating uncomplicated malaria in African children: a randomized trial. PLoS Med. 2011 Nov;8(11):e1001119. doi: 10.1371/journal.pmed.1001119. Epub 2011 Nov 8. PMID 22087077